CLINICAL TRIAL: NCT00879762
Title: Comparison of Safety and Immunogenicity of a High Dose (5 x 10^8 TCID50) and a Standard Dose (1 x 10^8 TCID50) of IMVAMUNE® in Healthy Vaccinia-Naive Individuals
Brief Title: High Dose IMVAMUNE® in Vaccinia-Naive Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 08-0040
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2012-01-26

CONDITIONS: Smallpox
Keywords: IMVAMUNE®; smallpox; vaccine
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: High Dose (Experimental): Single high dose of IMVAMUNE® (5x10^8 TCID50, consisting of two 0.5 mL injections) vaccine on Day 0 and a single saline placebo dose (single 0.5 mL injection) on Day 28 to match the two dose regimen of Group B.
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo
- Group B: Standard Dose (Active Comparator): Standard two dose regimen of IMVAMUNE® (1x10^8 TCID50) vaccine on Day 0 (consisting of 0.5 mL injection of vaccine and 0.5 mL injection of saline placebo) and Day 28 (single 0.5 mL injection of vaccine).
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo

INTERVENTIONS:
Biological: MVA Smallpox Vaccine — IMVAMUNE® Vaccinia Vaccine, undiluted, delivered by subcutaneous route on Day 0 at high dose 5×10^8 TCID50 (5×10^8 TCID50 per 1.0 mL dose - administered as 2 x 0.5 mL.
Other: Placebo — 0.5 mL injection of saline placebo administered with vaccine on Day 0 (Group B) or single saline placebo dose (single 0.5 mL injection) on Day 28 (Group A).

SUMMARY:
The purpose of this research is to compare the ability of a new investigational smallpox vaccine called IMVAMUNE® to produce a strong immune response against smallpox disease if given as one single, higher dose compared with two lower doses given one month apart. Another purpose of the study is to see how quickly someone might be protected against smallpox. Volunteers will be vaccinia-naïve adults age 18 and older (born after 1971) divided into 2 groups. Volunteers in Group A will receive a high dose of vaccine given in 2 shots on day 0 followed by a placebo (inactive substance) shot on day 28. Group B will receive the standard dose of vaccine and placebo given in 2 shots on day 0 followed by a standard dose shot on Day 28. Study participation will include 10 planned study visits over approximately 7 months.

DETAILED DESCRIPTION:
Despite the fact that the World Health Organization (WHO) officially declared smallpox to be eradicated, a new threat exists due to the potential use of variola virus as an agent for biological warfare and/or bio-terrorism. As a consequence, there is an urgent need for a safe and efficacious vaccine to protect the public against smallpox. To date, the majority of clinical studies with Modified Vaccinia Ankara (MVA) have studied a prime-boost vaccination regimen, with a dose of up to 1×10^8 tissue culture infectious dose 50 (TCID50) of MVA administered on Days 0 and 28. While this vaccination regimen induces a robust immune response that is protective in a variety of animal models and is appropriate for a pre-smallpox release scenario, in the event of a confirmed release of smallpox, a more rapid vaccination regimen that provides a protective immune response would be desirable. Ideally, at least short-term protection could be obtained with a single dose of vaccine. While a single dose of MVA at 1×10^8 TCID50, does induce an immune response in the majority of recipients, it is possible that a higher dose of MVA could provide a more rapid and/or stronger immune response relative to a single, standard 1×10^8 TCID50 dose of MVA. The goal of this study is to examine the kinetics and magnitude of the immune response of a single high dose of MVA (5×10^8 TCID50) relative to both a single and prime/boost regimen using the standard doses (1×10^8 TCID50) of MVA. This study will complement a current, ongoing study, DMID Protocol 06-0012, which is examining the immune response to compressed prime/boost dosing regimens of MVA administered at (1×10^8 TCID50). Upon the completion of these studies, clinical data will be generated which will inform policy makers about different options for post-event utilization of available smallpox vaccines. The study is designed as a randomized, non-placebo controlled, double blinded study containing two arms: Group A (N=45) will receive a single high dose of IMVAMUNE® (5x10^8 TCID50, consisting of two 0.5 mL injections) vaccine on Day 0 and a single saline placebo dose (single 0.5 mL injection) on Day 28 to match the two dose regimen of Group B. Group B (N=45) will receive a standard two dose regimen of IMVAMUNE® (1x10^8 TCID50) vaccine on Day 0 (consisting of 0.5 mL injection of vaccine and 0.5 mL injection of saline placebo) and Day 28 (single 0.5 mL injection of vaccine). Safety will be measured by assessment of adverse events for 28 days following the last vaccination (56 days following the initial vaccination for those subjects that fail to receive the second dose) and for serious adverse events at six months post the final vaccination, and reactogenicity to the vaccines for 15 days following each vaccination. Immunogenicity testing will include antibody testing [enzyme linked immunosorbent assay (ELISA) and plaque reduction neutralizing antibody titers (PRNT)] and cellular immune responses [(INF-gamma enzyme linked immunospot (ELISPOT)] following each vaccination and at six months post the final vaccination. In addition, ELISA responses, using MVA VR-1508 as the target antigen and PRNT using vaccinia WR (Western Reserve) as the target antigen will be explored. Participants will include 90 healthy, vaccinia-naïve adults, aged 18 and older (born after 1971). Study duration will be approximately 13 months (7 months/subject).

ELIGIBILITY:
Inclusion Criteria:

Prior to initial vaccination: -At least 18 years of age and born after 1971 -Read, sign, and date informed consent document -Available for follow-up for the planned duration of the study (six months after last immunization) -Acceptable medical history by screening evaluation and limited physical assessment -If the subject is female and of childbearing potential, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to vaccination -If the subject is female and of childbearing potential, she agrees to use acceptable contraception, and not become pregnant for 28 days following the last vaccination a. A woman is considered of childbearing potential unless post-menopausal (> 1 year) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy) b. Acceptable contraception methods are restricted to effective devices (IUDs, NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, abstinence from sexual intercourse with men (vaginal penetration by a penis, coitus), and monogamous relationship with a vasectomized partner. -Negative enzyme linked immunosorbent assay (ELISA) for human immunodeficiency virus (HIV) -Alanine aminotransferase (ALT) <1.25 times institutional upper limit of normal -Negative hepatitis B surface antigen and negative antibody to hepatitis C virus -Negative urine glucose and urine protein <1+ by dipstick or urinalysis -Adequate renal function is defined as a serum creatinine not exceeding the institution's upper limit of normal. - Electrocardiogram (ECG) in absence of clinical significance [e.g., complete left or right bundle branch block, incomplete left bundle branch block or sustained ventricular arrhythmia, or two premature ventricular contractions (PVC's) in a row, or sympathetic tonus (ST) elevation consistent with ischemia] -The following blood parameters: a. Hemoglobin equal or above the lower limit of institutional normal (sex specific); b. White blood cells greater than 2,500 and less than 11,000/mm^3; c. Platelets greater than or equal to 140,000/mm^3 -Weight greater than or equal to 110 pounds Inclusion Criteria that must be met prior to the second vaccination: -Acceptable medical history -ECG (obtained after Day 14 after first vaccination) in absence of clinical significance (e.g., complete left or right bundle branch block, incomplete left bundle branch block or sustained ventricular arrhythmia, or two PVC's in a row, or ST elevation consistent with ischemia) -If the subject is female and of childbearing potential, negative urine or serum pregnancy test within 24 hours prior to vaccination -If the subject is female and of childbearing potential, she agrees to use acceptable contraception, and not become pregnant for 28 days following the last vaccination a. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized b. Acceptable contraception methods are restricted to effective devices (IUDs, NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, and abstinence from sexual intercourse with men (vaginal penetration by a penis, coitus)

Exclusion Criteria:

Exclusion criteria that apply prior to the initial vaccination: -History of immunodeficiency -Typical vaccinia scar -Known or suspected history of smallpox vaccination including Modified Vaccinia Ankara (MVA) alone or as a vector as well as other investigational smallpox vaccine -Military service prior to 1991 or after January 2003 -Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease, diabetes mellitus, or moderate to severe kidney impairment -Malignancy not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site -Active autoimmune disease a. Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded -History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor -Systolic blood pressure >/= 150 mmHg or diastolic blood pressure >/= 100 mmHg. -Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp) NOTE that this criterion applies only to subjects 20 years of age and older and only if at least one of the following apply: a. Have smoked a cigarette in the past month, and/or b. Have hypertension (defined as systolic blood pressure >140 mm Hg) or are on antihypertensive medication, and/or c. Have a family history of coronary heart disease in male first-degree relative (father or brother) <55 years of age or a female first-degree relative (mother or sister) <65 years of age. -High-dose steroid use for greater than 2 weeks duration within three months prior to vaccination and current use of immunosuppressive medication. a. Corticosteroid nasal sprays are permissible b. Persons who are using a topical steroid can be enrolled after their therapy is completed c. Inhaled steroids for asthma are not permissible -Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol -Any history of illegal injection drug use -Receipt or planned receipt of inactivated vaccine from 14 days prior to the first vaccination through 14 days post second vaccination -Receipt or planned receipt of any other live attenuated vaccine within 30 days prior to the first vaccination through 30 days post second vaccination -Use of any other experimental agent within 30 days prior to vaccination and for the duration of the study -Receipt of blood products or immunoglobulin within six months prior to vaccination -Donation of a unit of blood within 56 days prior to vaccination or prior to Visit 9 -Acute febrile illness (greater than or equal to 100.5 degrees Fahrenheit) on the day of vaccination -Pregnant or lactating women -Eczema of any degree or history of eczema -People with active atopic dermatitis, active exfoliative skin disorders/conditions, current Varicella zoster, or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2×2 cm -Any condition that, in the opinion of the investigator, might interfere with study objectives -Known allergy to IMVAMUNE® vaccine -Known allergy to egg or aminoglycoside (including gentamicin) -Study personnel Exclusion criteria that apply prior to the second vaccination: -History of immunodeficiency -Known or suspected impairment of immunologic function including, but not limited to, clinically sig nificant liver disease, diabetes mellitus, or moderate to severe kidney impairment -Malignancy not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site -Active autoimmune disease a. Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded -History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor -Systolic blood pressure >/= 150 mmHg or diastolic blood pressure >/=100 mmHg -High-dose steroid use for greater than 2 weeks duration within three months prior to vaccination and current use of immunosuppressive medication. a. Corticosteroid nasal sprays are permissible b. Persons who are using a topical steroid can be enrolled after their therapy is completed c. Inhaled steroids for asthma are not permissible -Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol -Any history of illegal injection drug use -Receipt or planned receipt of inactivated vaccine from 14 days prior to vaccination through 14 days post second vaccination -Receipt or planned receipt of any other live attenuated vaccine from 30 days prior to vaccination through 30 days post second vaccination -Use of any other experimental agent within 30 days prior to vaccination and for the duration of the study -Receipt of blood products or immunoglobulin within six months prior to vaccination -Donation of a unit of blood within 56 days prior to vaccination or prior to Visit 9 -Acute febrile illness (greater than or equal to 100.4 degrees Fahrenheit) on the day of vaccination -Pregnant or lactating women -Eczema of any degree or history of eczema -People with active atopic dermatitis, active exfoliative skin disorders/conditions, current Varicella zoster, or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2×2 cm -Any condition that, in the opinion of the investigator, might interfere with study objectives -Known allergy to IMVAMUNE® vaccine -Known allergy to egg or aminoglycoside (including gentamicin)

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2009-05-29 (Actual); Primary Completion 2011-03-09 (Actual); Study Completion 2011-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included vaccinia-naïve adults aged greater than 18 years (and born after 1971). Participants were recruited from two sites within the United States. The first participant was enrolled on May 29, 2009, and the last participant was enrolled on August 16, 2010.
Groups:
- Group A: High Dose: Single high dose of IMVAMUNE® (5x10^8 TCID50, consisting of two 0.5 mL injections) vaccine on Day 0 and a single saline placebo dose (single 0.5 mL injection) on Day 28 to match the two dose regimen of Group B.
  IMVAMUNE® High Dose: IMVAMUNE® Vaccinia Vaccine, undiluted, delivered by subcutaneous route on Day 0 at high dose 5×10^8 TCID50 (5×10^8 TCID50 per 1.0 mL dose - administered as 2 x 0.5 mL.
  Placebo: 0.5 mL injection of saline placebo administered with vaccine on Day 0 (Group B) or single saline placebo dose (single 0.5 mL injection) on Day 28 (Group A).
- Group B: Standard Dose: Standard two dose regimen of IMVAMUNE® (1x10^8 TCID50) vaccine on Day 0 (consisting of 0.5 mL injection of vaccine and 0.5 mL injection of saline placebo) and Day 28 (single 0.5 mL injection of vaccine).
  Placebo: 0.5 mL injection of saline placebo administered with vaccine on Day 0 (Group B) or single saline placebo dose (single 0.5 mL injection) on Day 28 (Group A).
  IMVAMUNE® Standard Dose: IMVAMUNE® Vaccinia Vaccine delivered by subcutaneous (SC) route on Day 0 and 28 at standard dose (diluted with saline by study pharmacist to (1×10^8 tissue culture infectious dose 50 [TCID50] per 0.5 mL dose)
Period: Overall Study
Arm/Group | Group A: High Dose | Group B: Standard Dose
Started | 46 | 45
Completed | 43 | 44
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants. One participant in Group A was excluded because they received an incorrect dose for the first vaccination that did not correspond to either study group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: High Dose | Group B: Standard Dose | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (4.6) | 26.8 (4.8) | 26.8 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 42 | 42 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 41 | 39 | 80
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Seroconversion After One Vaccination Using Bavarian Nordic's (BN) Enzyme Linked Immunosorbent Assay (ELISA) in the Intent-to-Treat (ITT) Population
Description: Seroconversion is defined as a titer >= 50 or as a 2-fold or greater increase in titer from baseline if pre-vaccination titer was >= 50. Participants who did not seroconvert during the study were analyzed as right censored at the last sample collection date. Samples collected after the second vaccination were also analyzed as right censored.
Time Frame: Days 0, 4, 8, 14, 21, and 28 after first vaccination
Population: The ITT population includes all participants enrolled and randomized. Participants in this population are analyzed according to the group they were randomized to.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 46 | 45
days | 14 [13 to 14] | 14 [13 to 14]
Statistical Analysis 1: Comparison: Group A: High Dose vs Group B: Standard Dose; Null hypothesis: Median time to seroconversion among participants receiving one standard dose in Group B is 2.5-fold higher compared to participants receiving one high dose in Group A (hazard ratio = 2.5); Test type: Non-Inferiority — The non-inferiority margin is 2.5. Non-inferiority of Group B is concluded if the upper limit of the 95% confidence interval for the hazard ratio is less than 2.5; Hazard Ratio (HR) = 0.587, 95% CI 2-sided [0.398 to 0.868] — A survival analysis for interval censored data was performed to estimate the hazard ratio. The 95% CI for the hazard ratio was estimated using bootstrap

2. Primary Outcome: Time to Seroconversion After One Vaccination Using BN ELISA in the Per Protocol Population
Description: as for outcome 1
Time Frame: Days 0, 4, 8, 14, 21, and 28 after first vaccination
Population: The per protocol population includes all participants who received one dose of vaccine and contributed both pre- and post-vaccination blood samples for testing for which valid results were reported. One participant in Group A was additionally excluded due to receiving an incorrect dose for the first vaccination that did not correspond to either study group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 45 | 45
days | 14 [13 to 14] | 14 [13 to 14]
Statistical Analysis 1: Comparison: Group A: High Dose vs Group B: Standard Dose; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.583, 95% CI 2-sided [0.384 to 0.853] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Frequency of Serious Adverse Events (SAEs) Related to Vaccination
Description: The number of participants who experienced at least one SAE throughout the course of the study that was deemed related to the study vaccination. A SAE is defined as an AE meeting one of the following conditions:
  * Death during the study period (from first vaccine until end of surveillance period)
  * Life-threatening (defined as a participant at immediate risk of death at the time of the event)
  * Requires inpatient hospitalization or prolongation of existing hospitalization during the period of protocol-defined surveillance
  * Results in a congenital anomaly or birth defect
  * Results in a persistent or significant disability/incapacity
  * Severe adverse event associated with study product
Time Frame: Day 0 after first vaccination to study completion through Day 180 after second vaccination (Day 208 after first vaccination)
Population: The safety population includes all participants who received one dose of vaccine. One participant in Group A was additionally excluded due to receiving an incorrect dose for the first vaccination that did not correspond to either study group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 45 | 45
Participants | 0 | 0

4. Primary Outcome: Frequency of Non-Serious AEs Related to Vaccination
Description: The number of participants who experienced at least one unsolicited non-serious AE of any severity from Day 0 to 28 days post second vaccination (56 days post first vaccination) that was deemed related to the study vaccination.
Time Frame: Day 0 after first vaccination to Day 28 after second vaccination (Day 56 after first vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 45 | 45
Participants | 11 | 9

5. Primary Outcome: Frequency of Local Solicited Reactogenicity AEs for Subjective Symptoms
Description: Local solicited reactogenicity AEs were collected daily for 15 days post each vaccination using a memory aid. Local subjective events included pain at injection site, itchiness at injection site, underarm pain, and underarm swelling and were graded on a scale of Grade 0 (None), Grade 1 (Mild), Grade 2 (Moderate), and Grade 3 (Severe).
Time Frame: Day 0 through Day 15 after first vaccination; Day 0 through Day 15 after second vaccination (Day 28 through Day 43 after first vaccination)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 45 | 45
Participants
  Post Vaccination 1 (Day 0 through Day 15): number analyzed (Participants) | 45 | 44
  Post Vaccination 1 (Day 0 through Day 15) | 41 | 34
  Post Vaccination 2 (Day 28 through Day 43): number analyzed (Participants) | 43 | 41
  Post Vaccination 2 (Day 28 through Day 43) | 7 | 33

6. Primary Outcome: Frequency of Local Solicited Reactogenicity AEs for Measured Symptoms
Description: Local solicited reactogenicity AEs were collected daily for 15 days post each vaccination using a memory aid. Local measured events included erythema and induration at the vaccination site and were measured in millimeters.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 45 | 45
Participants
  Post Vaccination 1 (Day 0 through Day 15): number analyzed (Participants) | 45 | 44
  Post Vaccination 1 (Day 0 through Day 15) | 26 | 22
  Post Vaccination 2 (Day 28 to Day 43): number analyzed (Participants) | 43 | 41
  Post Vaccination 2 (Day 28 to Day 43) | 3 | 20

7. Primary Outcome: Frequency of Systemic Solicited Reactogenicity AEs
Description: Systemic solicited reactogenicity AEs were collected daily for 15 days post each vaccination using a memory aid. Systemic events included muscle aches, chills, headache, nausea, feeling tired, change in appetite, joint pain, and elevated oral temperature. Events were graded on a scale of Grade 0 (None), Grade 1 (Mild), Grade 2 (Moderate), and Grade 3 (Severe).
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 45 | 45
Participants
  Post Vaccination 1 (Day 0 through Day 15) | 27 | 19
  Post Vaccination 2 (Day 28 to Day 43): number analyzed (Participants) | 43 | 42
  Post Vaccination 2 (Day 28 to Day 43) | 7 | 11

8. Secondary Outcome: Peak Titer of Saint Louis University's (SLU) Plaque Reduction Neutralizing Antibody Titer (PRNT) Assay After First Vaccination in the ITT Population
Description: The peak PRNT is defined as the largest titer among all available measurements post-first vaccination but prior to the second vaccination. Means and corresponding standard errors are calculated on the log2.5 scale.
Time Frame: Days 4, 8, 14, 21, and 28 after first vaccination
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log2.5 of titer
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 46 | 45
log2.5 of titer | 4.94 (0.19) | 4.56 (0.23)
Statistical Analysis 1: Comparison: Group A: High Dose vs Group B: Standard Dose; Null hypothesis: The mean difference in log2.5 transformed peak titers between Group A and Group B >= 1; Test type: Non-Inferiority — The non-inferiority margin is 1. Non-inferiority of Group B is concluded if the upper limit of the 95% confidence interval for the mean difference in the log2.5 transformed peak titers between groups is less than 1; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.20 to 0.97] — Estimate and corresponding 95% confidence interval are calculated on the log2.5 scale

9. Secondary Outcome: Peak Titer of SLU PRNT Assay After First Vaccination in the Per Protocol Population
Description: as for outcome 8
Time Frame: Days 4, 8, 14, 21, and 28 after first vaccination
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log2.5 of titer
Arm/Group | Group A: High Dose | Group B: Standard Dose
Number analyzed (Participants) | 45 | 45
log2.5 of titer | 4.98 (0.19) | 4.56 (0.23)
Statistical Analysis 1: Comparison: Group A: High Dose vs Group B: Standard Dose; Null hypothesis: The mean difference in log2.5 transformed peak titers between Group A and Group B >= 1; Test type: Non-Inferiority — [test comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.17 to 1.00] — Estimate and corresponding 95% confidence interval are calculated on the log2.5 scale

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected daily for 15 days post each vaccination. Unsolicited AEs were reported from the first vaccination through 28 days post second vaccination (56 days post first vaccination). SAEs were reported from the first vaccination to study completion (Day 208 post first vaccination).
Description: AEs are presented by actual study product received. One participant in Group A was excluded due to receiving an incorrect dose for the first vaccination that did not correspond to either study group.
Arm/Group | Group A: High Dose | Group B: Standard Dose
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 45/45 | 43/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: High Dose (N=45) | Group B: Standard Dose (N=45)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vaccination site discolouration (General disorders) | 3 (3) | 5 (6)
Vaccination site haematoma (General disorders) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (5)
Axillary pain (General disorders) | 5 (5) | 9 (11)
Chills (General disorders) | 5 (5) | 2 (2)
Fatigue (General disorders) | 15 (20) | 11 (13)
Underarm swelling (General disorders) | 3 (3) | 4 (5)
Vaccination site erythema (General disorders) | 23 (25) | 30 (43)
Vaccination site pain (General disorders) | 40 (45) | 39 (68)
Vaccination site pruritus (General disorders) | 10 (10) | 10 (14)
Vaccination site swelling (General disorders) | 22 (22) | 27 (36)
Appetite disorder (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (18) | 10 (12)
Headache (Nervous system disorders) | 17 (21) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less